CLINICAL TRIAL: NCT01696110
Title: Bivalirudin in Acute Myocardial Infarction vs Glycoprotein IIb/IIIa and Heparin Undergoing Angioplasty (BRIGHT):a Randomised Controlled Trial
Brief Title: BivaliRudin in Acute Myocardial Infarction vs Glycoprotein IIb/IIIa and Heparin :a Randomised Controlled Trial.
Acronym: BRIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, director of the department of cardiology, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYNH20120001; 2011BAI11B07 (Other Grant/Funding Number: China National Science and Technology support project plan)
Record Dates: First submitted 2012-08-22; First posted 2012-09-28 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: Bivalirudin; Acute myocardial infarction; percutaneous transluminal coronary angioplasty
MeSH Terms: interventions — bivalirudin; Heparin; Tirofiban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bivalirudin (Experimental): Bivalirudin will be started in the cath lab, 0.75 mg/kg intravenous bolus followed by 1.75 mg/kg per h infusion; if ACT<225s 5min after bolus, an additional dose of 0.3mg/kg bolus should be given. After procedure, a prolonged infusion (1.75mg/kg per h) will be given for at least 30 min (totally no more than 4 h) followed by a reduced dose infusion (0.2mg/kg per h) up to 20 h.
  Interventions: Drug: Bivalirudin
- Heparin monotherapy (Active Comparator): 100 IU/kg intravenous bolus. If ACT <225s 5 min after bolus injection, additional dose of heparin (20U/kg) will be given.
  Interventions: Drug: heparin
- heparin plus tirofiban (Active Comparator): heparin 60 IU/kg intravenous bolus and Tirofiban: 10μg/kg intravenous bolus followed by 0.15μg/kg per min infusion for up to 36h.
  Interventions: Drug: heparin; Drug: heparin plus tirofiban

INTERVENTIONS:
Drug: Bivalirudin — Patients would be given anticoagulant therapy with bivalirudin in acute myocardial infarction during emergency PCI operation.
  Other Names: Taijianing
  Arms: Bivalirudin
Drug: heparin — heparin monotherapy
  Arms: Heparin monotherapy; heparin plus tirofiban
Drug: heparin plus tirofiban — combined use of heparin and tirofiban during PCI
  Other Names: brand name of tirofiban: Xinweining
  Arms: heparin plus tirofiban

SUMMARY:
The study would enrolled a total of 2100 AMI patients undergoing PCI to one of three antithrombotic regimens: bivalirudin alone, or unfractionated heparin alone, or unfractionated heparin plus a glycoprotein IIb/IIIa inhibitor.

All enrolled patients would be followed-up to 30 days, 6 months, and 1 year. The purpose of the study is to evaluate the efficacy and safety of bivalirudin in AMI patients with DES.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, active drug controlled multicenter clinical research and the study would enrolled a total of 2100 AMI patients undergoing percutaneous coronary intervention (PCI) to one of three antithrombotic regimens: bivalirudin alone, or unfractionated heparin alone, or unfractionated heparin plus a glycoprotein IIb/IIIa inhibitor. All enrolled patients would be followed-up to 30 days, 6 months, and 1 year. The purpose of the study is to evaluate the efficacy and safety of bivalirudin in AMI patients with DES.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old
2. Planned emergency PCI for acute myocardial infarction (STEMI or NSTEMI) Symptom onset within 12h for STEMI (or within 24 h for patients have unrelieved chest pain, continuous ST elevation or new developed LBBB) Symptom onset within 72h for NSTEMI
3. Avoid to undergoing revascularization for non-culprit vessels within 30 days after index procedure.
4. Provide written informed consent.

Exclusion Criteria:

1. Unsuitable for PCI; treatment by thrombolysis within 72 hours of acute ST-elevation myocardial infarction; left main coronary artery disease; cardiogenic shock.
2. Any anticoagulant agents were used 48 h before randomization.
3. Active bleeding or bleeding constitution, bleeding tendency, including the recent retina or vitreous hemorrhage (1 months), GI or urinary tract hemorrhage (3 months), cerebral hemorrhage (6 months) or cerebral infarction history (3 months), etc.;
4. Other disease may lead to vascular lesions and secondary bleeding factors (such as active gastric ulcer, active ulcerative colitis, intracranial aneurysm, etc.),
5. Deep puncture or major surgery (including eye or brain surgery) within 1 month.
6. Suspicious aortic dissection, pericarditis and subacute bacterial endocarditis.
7. Untreated or uncontrolled hypertension > 180/110 mmHg.
8. Hemoglobin < 100 g/L or platelet count < 100 * 109 / L.
9. Elevated AST, ALT level higher than three times of the normal upper limit.
10. severe renal insufficiency (eGFR < 30 mL/min / 1.73 m2).
11. Heparin induced thrombocytopenia.
12. Known allergy to the study drugs and instruments (UFH, bivalirudin, aspirin and clopidogrel, stainless steel, contrast agents, etc.), or those allergic constitution.
13. Pregnancy or lactation.
14. Researchers think that doesn't fit to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2194 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Net Adverse Clinical Events | 30 days
  A composite of all cause death, reinfarction, urgent target vessel revascularization, stroke and any bleedings

SECONDARY OUTCOMES:
Net adverse clinical events | 1 year
  a composite of all cause death, any myocardial infarction, any target vessel revascularization, stroke or any bleedings
any bleedings (BARC class) | 30 day
  including all BARC class (class 1-5)
Major adverse cardiac and cerebral events (MACCE) | 30 days and 1 year
  a composite of all cause death, reinfarction, target vessel revascularization or stroke

OTHER OUTCOMES:
Thrombocytopenia | 30 days
  Defined as a decrease of platelet count of more than 50% or more than 150000 platelet/mm3 compared with baseline within 24h after study drug administration
stent thrombosis | 30 days and 1 year
  by ARC definition

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — Shenyang Northern Hospital,China
Locations (81):
- China (81):
  - 1 st Hosp. of Anhui Med Univ., Hefei, Anhui
  - Anhui Provincial Hosp., Hefei, Anhui
  - 3rd Hosp. of Beijing Univ., Beijing, Beijing Municipality
  - Beijing Anzhen Hosp., Beijing, Beijing Municipality
  - Beijing CAPF General Hosp., Beijing, Beijing Municipality
  - Beijing Chaoyang Hosp., Beijing, Beijing Municipality
  - Beijing Friendship Hosp., Beijing, Beijing Municipality
  - Beijing General Hosp. of PLA, Beijing, Beijing Municipality
  - Beijing Hosp., Beijing, Beijing Municipality
  - Beijing Luhe Hosp., Beijing, Beijing Municipality
  - General Hosp of PLA (1), Beijing, Beijing Municipality
  - General Hosp. of PLA(2), Beijing, Beijing Municipality
  - Navy General Hosp. of PLA, Beijing, Beijing Municipality
  - No.304 Hosp. of PLA, Beijing, Beijing Municipality
  - No.306 Hosp. of PLA, Beijing, Beijing Municipality
  - Peking Univ. First Hosp., Beijing, Beijing Municipality
  - The 2nd artillery general Hosp. of PLA, Beijing, Beijing Municipality
  - Chongqing Daping Hosp., Chongqing, Chongqing Municipality
  - Fujian Med Univ. Uion Hosp., Fuzhou, Fujian
  - 1 st Hosp. of Lanzhou Univ., Lanzhou, Gansu
  - Lanzhou General Hosp. of PLA, Lanzhou, Gansu
  - 1 st Hosp. of Guangzhou MU, Guangzhou, Guangdong
  - 1st Hosp. of Zhongshan MU, Guangzhou, Guangdong
  - Guangdong General Hosp., Guangzhou, Guangdong
  - Guangzhou General Hosp. of PLA, Guangzhou, Guangdong
  - 1 st Hosp. of Guangxi Med Univ., Nanning, Guangxi
  - No.252 Hosp. of PLA, Baoding, Hebei
  - Cangzhou Centeral Hosp., Cangzhou, Hebei
  - Qinhuangdao No.1 Hosp., Qinhuangdao, Hebei
  - Hebei General Hosp., Shijiazhuang, Hebei
  - Shijiazhuang Peace Hosp., Shijiazhuang, Hebei
  - Tangshan Gongren Hosp., Tangshan, Hebei
  - Daqing General Hosp. of OF., Daqing, Heilongjiang
  - No.152 Hosp., Pingdingshan, Henan
  - Wuhan Asican Heart Hosp., Wuhan, Hubei
  - Wuhan General Hosp of PLA, Wuhan, Hubei
  - Nanjing First Hosp., Nanjing, Jiangsu
  - Xuzhou Med Col. Affiliated Hosp., Xuzhou, Jiangsu
  - Xuzhou No.4 Hosp., Xuzhou, Jiangsu
  - 2 nd Hosp. of Nanchang Univ., Nanchang, Jiangxi
  - 1st Hosp of Jilin Univ., Changchun, Jilin
  - 2nd Hosp of Jilin Univ., Changchun, Jilin
  - 3rd Hosp of Jilin Univ., Changchun, Jilin
  - Meihekou Central Hosp., Meihekou, Jilin
  - Dalian Zhongshan Hosp., Dalian, Liaoning
  - No.210 Hosp of PLA, Dalian, Liaoning
  - No.313 Hosp. of PLA, Huludao, Liaoning
  - 1st Hosp. of Liaoning MC, Jinzhou, Liaoning
  - 3 rd Hosp. of Liaoning Med Col., Jinzhou, Liaoning
  - No.463 Hosp of PLA, Shenyang, Liaoning
  - Shenzhou Hosp. of SMC, Shenyang, Liaoning
  - Yingkou Centeral Hosp., Yingkou, Liaoning
  - General Hosp. of Ningxia MU, Yinchuan, Ningxia
  - Ji'nan General Hosp. of PLA, Ji'nan, Shandong
  - Affiliated Hosp. of Jining MC, Jining, Shandong
  - Taian Central Hosp., Taian, Shandong
  - Yantaishan Hosp., Yantai, Shandong
  - No. 148 Hosp., Zibo, Shandong
  - Huashan Hosp., Shanghai, Shanghai Municipality
  - Shanghai jingan people's hosp., Shanghai, Shanghai Municipality
  - Shanghai Renji Hosp., Shanghai, Shanghai Municipality
  - 1st Hosp. of Shanxi Med Univ., Taiyuan, Shanxi
  - Shanxi Cardiovascular Hosp., Taiyuan, Shanxi
  - Taiyuan Central Hosp., Taiyuan, Shanxi
  - 2 nd Hosp. of Xi'an Med Col., Xi’an, Shanxi
  - Shanxi General Hosp. of CAPF, Xi’an, Shanxi
  - Shanxi General Hosp., Xi’an, Shanxi
  - Tangdu Hosp., Xi’an, Shanxi
  - Xijing Hosp., Xi’an, Shanxi
  - Yanan Univ. affiliated Hosp., Yanan, Shanxi
  - Yuncheng Central Hosp., Yuncheng, Shanxi
  - Chengdu General Hosp. of PLA, Chengdu, Sichuan
  - Chengdu No.2 Hosp., Chengdu, Sichuan
  - No.254 Hosp. of PLA, Tianjin, Tianjin Municipality
  - Tianjin CAPF Hosp., Tianjin, Tianjin Municipality
  - Tianjin Chest Hosp., Tianjin, Tianjin Municipality
  - Tianjin No.3 Hosp., Tianjin, Tianjin Municipality
  - Tianjin People's Hosp., Tianjin, Tianjin Municipality
  - Kunming General Hosp. of PLA, Kunming, Yunnan
  - 2nd Hosp. of Zhejiang Univ., Hangzhou, Zhejiang
  - Zhejiang Hosp., Hangzhou, Zhejiang

REFERENCES:
- [Derived] Liang Z, Li Y, Wang J, Wang D, Wang S, Ma L, Liu H, Yang L, Stone GW, Han Y. The safety and effectiveness of bivalirudin in female patients with acute myocardial infarction undergoing primary angioplasty: A subgroup analysis of the BRIGHT trial. Catheter Cardiovasc Interv. 2016 Mar;87 Suppl 1:608-15. doi: 10.1002/ccd.26407. Epub 2016 Jan 13. PMID 26762481
- [Derived] Han Y, Guo J, Zheng Y, Zang H, Su X, Wang Y, Chen S, Jiang T, Yang P, Chen J, Jiang D, Jing Q, Liang Z, Liu H, Zhao X, Li J, Li Y, Xu B, Stone GW; BRIGHT Investigators. Bivalirudin vs heparin with or without tirofiban during primary percutaneous coronary intervention in acute myocardial infarction: the BRIGHT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1336-46. doi: 10.1001/jama.2015.2323. PMID 25775052